CLINICAL TRIAL: NCT07382531
Title: An Open-label, Dose-escalation Phase Ib/II Clinical Trial of Intratumoral Injection of OH2 Injection in Combination With BS006 Injection for the Treatment of Advanced Solid Tumors.
Brief Title: OH2 Injection in Combination With BS006 Injection for Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Binhui Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BS008-001
Record Dates: First submitted 2026-01-27; First posted 2026-02-02 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Solid Tumor

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- OH2+BS006 (Experimental): The administration method consists of sequential intratumoral injections of OH2 and BS006 at an equal volume ratio. Administration occurs once every 2 weeks (Q2W) until the investigator determines that the subject no longer derives clinical benefit and exhibits significant clinical disease progression (radiographic progression is not a mandatory criterion for treatment discontinuation), or until the treatment is no longer tolerated, or the clinical trial concludes. For each administration, subjects may receive a maximum of 6 mL each of OH2 Injection and BS006 Injection.
  Interventions: Biological: OH2+BS006

INTERVENTIONS:
Biological: OH2+BS006 — Patients received biweekly sequential intratumoral injections of OH2 (fixed dose: 10⁷ CCID₅₀/mL) followed by BS006 (dose escalation: 10⁶-10⁷ CCID₅₀/mL), with identical volumes being injected at the same lesion.

SUMMARY:
BS008-001 is a multicenter, open-label phase Ib /II trial in heavily pre-treated patients with advanced solid tumors. Patients received biweekly sequential intratumoral injections of OH2 (fixed dose: 10⁷ CCID₅₀/mL) followed by BS006 (dose escalation: 10⁶-10⁷ CCID₅₀/mL), with identical volumes being injected at the same lesion. The primary endpoint is safety and tolerability; secondary endpoints included efficacy outcomes assessed by RECIST 1.1/iRECIST.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients with unresectable stage III or IV malignant tumors confirmed by pathology and/or cytology; such as malignant melanoma, head and neck tumors, soft tissue sarcoma, liver tumors (primary hepatocellular carcinoma or liver metastases), biliary tract tumors, pancreatic cancer, esophageal cancer, gastric cancer, etc.
* 2. Lack of standard effective treatment options, or failure of or relapse after standard treatments.
* 3.Male or female patients aged 18-75 years (inclusive); Eastern Cooperative Oncology Group (ECOG) performance status score of 0-1; expected survival of more than 3 months.
* 4. At least 4 weeks have elapsed since completion of prior antitumor therapies (including endocrine therapy, chemotherapy/radiotherapy, and targeted therapy) (except radiotherapy for bone metastases); for patients treated with nitrosoureas or mitomycin, at least 6 weeks since discontinuation; and recovery from prior treatment-related adverse effects to Grade 1 or lower.
* 5. Patients who have undergone major surgery must be at least 4 weeks post-operation.
* 6. According to RECIST 1.1 criteria, at least one measurable target lesion is required, with a lesion suitable for intratumoral injection. A measurable tumor lesion is defined as having a longest diameter ≥10 mm with a scan slice thickness ≤5.0 mm; for lymph node lesions, a short-axis diameter ≥15 mm.
* 7. No severe dysfunction of major organs.
* 8. Laboratory tests:

  1. White Blood Cell (WBC) ≥3.0×10⁹/L, Absolute Neutrophil Count (ANC) ≥2.0×10⁹/L, Hemoglobin (Hb) ≥90 g/L; Platelet (PLT) ≥100×10⁹/L; absolute lymphocyte count (ALC)≥0.8×10⁹/L;
  2. Blood urea nitrogen (BUN) and serum creatinine ≤1.5× the upper limit of normal (ULN);
  3. Total bilirubin (TBIL) ≤1.5× ULN (for patients with hepatic involvement, TBIL ≤3× ULN);
  4. Alanine Aminotransferase (ALT) and Aspartate Aminotransferase (AST) ≤2.5× ULN; for patients with liver metastases, ≤5× ULN;
  5. Normal coagulation function (Prothrombin Time, APTT, and Thrombin Time ≤1.5× ULN).
* 9. Female subjects and their partners must use effective contraception during treatment and for 3 months after treatment.
* 10. Subjects with genital herpes must have completed herpes resolution for at least 3 months.
* 11. Voluntary signing of the informed consent form, with expected good compliance.

Exclusion Criteria:

* 1. Concomitant serious medical diseases, including uncontrolled diabetes, severe infections, or active gastrointestinal ulcers.
* 2. Presence of clinically significant cardiovascular or cerebrovascular disease, including:

  1. Severe or uncontrolled heart disease requiring treatment, congestive heart failure classified as New York Heart Association (NYHA) class III or IV, unstable angina not controlled by medication, a history of myocardial infarction within the past 6 months, Corrected QT Interval (QTc) on Electrocardiogram (ECG) ≥450 ms in males or ≥470 ms in females, or severe arrhythmias requiring drug treatment (excluding atrial fibrillation or paroxysmal supraventricular tachycardia);
  2. Placement of a cardiac stent within the past 6 months;
  3. Inadequately controlled hypertension, defined as systolic blood pressure ≥160 mmHg and/or diastolic blood pressure ≥100 mmHg.
* 3.Uncontrolled primary brain tumors or brain metastases.
* 4. Bone metastases (except for bone metastases that are stable and controlled after treatment), or the presence of active, clinically symptomatic brain metastases.
* 5. Active autoimmune diseases requiring systemic treatment within the past 2 years (including but not limited to rheumatoid arthritis, systemic lupus erythematosus, Sjögren's syndrome, etc., such as the use of disease-modifying drugs, corticosteroids, or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiological corticosteroid replacement therapy for renal or pituitary insufficiency) is not considered a systemic treatment.
* 6. History of immunodeficiency (HIV antibody-positive), or other acquired or congenital immunodeficiency diseases, or a history of organ transplantation.
* 7. Uncontrolled psychiatric disorders or infectious diseases. Lesions that do not meet the volume requirements for intratumoral injection.
* 8. Patients with active hepatitis B or hepatitis C infection: those who are HBsAg-positive or HBcAb-positive with detectable HBV DNA copies (lower limit of quantification: 500 IU/mL); HBV DNA testing is mandatory at screening for such patients. Patients with a positive anti-HCV antibody test are eligible only if HCV RNA PCR testing is negative.
* 9. Positive HIV test result.
* 10. Presence of active tuberculosis infection or other infectious diseases requiring systemic treatment.
* 11. Large amounts of pleural effusion or ascites accompanied by clinical symptoms or requiring symptomatic treatment.
* 12. Pregnant or breastfeeding women.
* 13. Use of, or ongoing treatment with, other investigational drugs or antiviral therapies within 4 weeks prior to treatment, except that patients with chronic hepatitis B receiving continuous treatment may use entecavir, tenofovir disoproxil fumarate, or adefovir dipivoxil.
* 14. Participation in another clinical study within the past 4 weeks.
* 15. Known allergy to herpes viruses or any components of the study drug.
* 16. Any other condition that, in the investigator's judgment, makes the patient unsuitable for participation in this trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-09-07 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of AE (Adverse Event) and SAE (Serious Adverse Event) | Through study completion, six months after the last administration of the study drug to the last enrolled subject.
  Toxic reactions according to the NCI-CTCAE 5.0 grading standard that occur within 3 weeks from the first administration, are judged to be drug-related by the investigator, and meet the non-hematological toxicity and hematological toxicity conditions specified in the clinical protocol
DLTs (Dose Limiting Toxicity) | 4 weeks from the first administration
  Toxic reactions according to the NCI-CTCAE 5.0 grading standard that occur within 4 weeks from the first administration, are judged to be drug-related by the investigator, and meet the non-hematological toxicity and hematological toxicity conditions specified in the clinical protocol
MTD | Through study completion, six months after the last administration of the study drug to the last enrolled subject.
  If ≥2/6 subjects developed DLT, the previous dose group was MTD

SECONDARY OUTCOMES:
ORR/iORR | Through study completion, six months after the last administration of the study drug to the last enrolled subject.
  Tumor response will be assessed according to RECIST 1.1 and iRECIST criteria. Descriptive statistics will be used to calculate the number and proportion of subjects achieving objective response (CR/iCR + PR/iPR) at each evaluation time point.
DOR/iDOR | Through study completion, six months after the last administration of the study drug to the last enrolled subject.
  The Kaplan-Meier method will be used to estimate the median duration of response (DoR).
PFS/iPFS | Through study completion, six months after the last administration of the study drug to the last enrolled subject.
  The Kaplan-Meier method will be used to estimate the median progression-free survival.
DCR/iDCR | Through study completion, six months after the last administration of the study drug to the last enrolled subject.
  umor assessments will be performed according to RECIST 1.1 and iRECIST criteria. Descriptive statistics will be used to calculate the number and proportion of subjects achieving complete response (CR/iCR), partial response (PR/iPR), and stable disease (SD/iSD) at each assessment time point.
OS | Through study completion, six months after the last administration of the study drug to the last enrolled subject.
  The Kaplan-Meier method will be used to estimate the median overall survival (OS).

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongnan Hospital of Wuhan University, Wuhan, Hubei, China